CLINICAL TRIAL: NCT01792375
Title: Concurrent Membrane Sweeping With Dinoprostone Versus Dinoprostone in Labor Induction of Nulliparas at Term With an Unfavorable Cervix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWP_PG_Null
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2016-10

CONDITIONS: Nulliparous Women Who Scheduled for Labor Induction
Keywords: Cervical ripening; Dinoprostone; Labor induction; Membrane sweeping; Nulliparous women; Trial
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Concurrent membrane sweeping with Dinoprostone (Active Comparator)
  Interventions: Procedure: Concurrent membrane sweeping with Dinoprostone
- Dinoprostone (Active Comparator)
  Interventions: Drug: 10mg Dinoprostone vaginal insert

INTERVENTIONS:
Procedure: Concurrent membrane sweeping with Dinoprostone — Women assigned to "Sweep" had their cervix swept by inserting the examining finger as high as possible past the internal cervical os, immediately followed by the placement of a 10mg Dinoprostone vaginal insert in the posterior fornix.
  Arms: Concurrent membrane sweeping with Dinoprostone
Drug: 10mg Dinoprostone vaginal insert — For women assigned to "No sweep": The only 10mg Dinoprostone vaginal insert were placed in the posterior fornix for cervical ripening
  Arms: Dinoprostone

SUMMARY:
To compare concurrent membrane sweeping with dinoprostone versus dinoprostone in labor induction for nulliparas at term with an unfavorable cervix

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* Nulliparous women
* gestational age >=37.0 weeks
* Bishop score <=6
* intact amniotic membrane
* absence of labor
* live fetus with vertex presentation
* no previous uterine surgical procedure

Exclusion Criteria:

* Multiple pregnancy
* Placenta previa

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2013-02; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Vaginal delivery within 24 hours | Twenty-four hours of initiating intervention (i.e. membrane sweeping or PG) on the first day of induction
  Vaginal delivery within 24 hours is defined as vaginal delivery after 24 hours of initiating intervention (i.e. concurrent membrane sweeping with dinoprostone or only dinoprostone) on the first day of induction.

SECONDARY OUTCOMES:
Cervical change in the bishop scores and cervical lengths | Initiation of oxytocin after removing dinoprostone vaginal insert
  1. Cervical change based on the bishop score and cervical length induced by two cervical ripening methods(concurrent membrane sweeping with dinoprostone vs. dinoprostone)
  2. Incidence of cesarean delivery
  3. Successful labor induction (defined as an ability to achieve the active phase of labor corresponding to a cervical dilatation of >=4cm).
  4. The interval from start of oxytocin to delivery
  5. Incidence of rupture of membranes
  6. Incidences of vaginal bleeding and fever

CONTACTS AND LOCATIONS:
Overall Officials: Kyo Hoon Park, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Department of Obstetrics and Gynecology Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea